CLINICAL TRIAL: NCT06973473
Title: Aprospective,Randomized,Comparative Clinical Trial of Combination Therapy of Imiquimod 5%Cream and Cryotherapy vs Monotherapy for Common Warts.
Brief Title: Combination Therapy of Imiquimod 5%Cream and Cryotherapy vs Monotherapy for Common Warts:Randomized Comparative Trial.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa yahia mohamed hassan, candidate, Assiut University
Other Study IDs: Treatment of common warts
Record Dates: First submitted 2025-04-29; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the clinical efficacy and safety of topical imiquimod 5% cream combined with cryotherapy versus either of theme alone for the treatment of common warts by clinical and dermoscopic assessments.

DETAILED DESCRIPTION:
Topical Imiquimod 5% cream Combined with Cryotherapy Versus either of them alone in Treatment of Common Warts: A prospective Randomized Comparative Trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with common warts diagnosed clinically and by dermoscopy.
* Patients older than 18years old.

Exclusion Criteria:

* Pregnancy and lactation.
* Immunosuppression or being under any kind of treatment causing
* absolute or relative immunosuppression.
* Patients with chronic systemic diseases.
* All cases of bleeding tendency or using anticoagulants.
* Concurrent use of systemic or topical treatments of warts in the last 4 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: - study population age older than 18years
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete clearance rate of common warts. | 12 weeks
  Assessment of complete warts clearance rate at 12weeks to evaluate the efficacy of combination therapy ( imiquimod5%cream+cryotherapy ) compared to topical imiquimod5%cream alone or cryotherapy alone in patients with common wart.

IPD SHARING:
Plan to Share IPD: No